CLINICAL TRIAL: NCT00965029
Title: Spirometry in Mechanically Ventilated COPD Patients: Correlation of Lung Function Tests to Successful Weaning From Mechanical Ventilation
Brief Title: Spirometry in Mechanically Ventilated Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Arie Soroksky, M.D., General ICU, Assaf Harofe Medical Center, Zerifin 70300, Israel
Other Study IDs: 101/09
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2009-08

CONDITIONS: COPD
Keywords: COPD; Spirometry; Weaning
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with COPD who deteriorate to Respiratory Failure pose a challenge to the intensivist both in ventilating an obstructed patient and in weaning from mechanical ventilation.

Currently there are no accepted extubation criteria in COPD patients that could predict successful weaning from mechanical ventilation. In this study we will attempt to correlate spirometric data to eventual weaning from mechanical ventilation.

DETAILED DESCRIPTION:
COPD patients who deteriorate to Respiratory Failure will be recruited. Sedation will be interrupted daily, and each day once the patient is awake and cooperative, spirometry will be performed. FEV1 and FVC will be recorded and later correlated to eventual rate of successful extubation.

ELIGIBILITY:
Inclusion Criteria:

* >18
* Mechanically ventilated due to COPD exacerbation

Exclusion Criteria:

* decreased level of consciousness
* uncooperative patient
* Bronchial asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients with respiratory failure due to COPD exacerbation, and on mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Arie Soroksky, MD, Principal Investigator — General ICU, Assaf Harofe MC, Zerifin, Israel
Locations (1):
- Arie Soroksky, Beer Yaakov, Zerifin, Israel